CLINICAL TRIAL: NCT03211039
Title: Prenatal Precision Medicine (NSIGHT2): A Randomized, Blinded, Prospective Study of the Clinical Utility of Rapid Genomic Sequencing for Infants in the Acute-care Setting
Brief Title: Perinatal Precision Medicine
Acronym: NSIGHT2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rady Pediatric Genomics & Systems Medicine Institute (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Stephen F. Kingsmore, President and CEO, Rady Pediatric Genomics & Systems Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 161983; U19HD077693 (NIH)
Record Dates: First submitted 2017-05-24; First posted 2017-07-07 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Genetic Diseases; Genetic Syndrome; Mendelian Disorders
Keywords: Neonate; Genomic Medicine; Rapid Precision Medicine; Rapid Whole Genome Sequencing; Diagnosis; Infant; Intensive care unit; clinical trial; Rapid Whole Exome Sequencing; Single locus disease; Ultra-rapid whole genome sequencing; Clinical Utility
MeSH Terms: conditions — Genetic Diseases, Inborn; Disease

STUDY DESIGN:
Intervention Model Description: The initial symptom-driven analysis will be conducted on the patient's (NICU infants) sample only (singleton analysis). Patients will be randomized to receive either whole genome sequencing or whole exome sequencing. If a diagnosis is not found promptly (within 24 hours) via singleton analysis, sequential analysis of the family (or any combination of parents and/or other family members) will be analyzed using the same technology that the patient was randomized to receive.
  The study includes parental and physician questionnaires to understand perceptions regarding testing. There is no randomization of parents or physicians nor a requirement to respond to the questionnaires for the patient (NICU infant) to participate in the study.
  Enrollment: 213 patients (NICU infants)
Who Masked: Participant
Masking Description: Patients (NICU infants) and their parents, the patient's providers, and the enrollment staff will be blinded to the randomization arm they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Whole Genome Sequencing (Other): Genetic test that looks at all coding and non-coding areas of the genome
  Interventions: Genetic: Genomic sequencing and molecular diagnostic results, if any.
- Whole Exome Sequencing (Other): Genetic test that looks at all coding areas of the genome
  Interventions: Genetic: Genomic sequencing and molecular diagnostic results, if any.

INTERVENTIONS:
Genetic: Genomic sequencing and molecular diagnostic results, if any. — Patients and their families will be randomized to either receive whole genome sequencing or whole exome sequencing.

SUMMARY:
This study will seek to determine if rapid genomic sequencing improves outcomes for acutely ill infants. The investigator will enroll up to 1,000 acutely ill infants in a prospective, randomized, blinded study to either rapid Whole Genome Sequencing (WGS) or rapid Whole Exome Sequencing (WES, which is 2% of the genome and ~4-fold less expensive). 213 infants were actually enrolled. Outcomes will be measured both by objective clinical measures and family perceptions (patient/family centered outcomes). Primary analysis of WGS or WES will be in infants alone. Secondary analysis, in infants who do not receive a diagnosis, will be of families - ideally trios (mother, father, and affected infant), which is ~2-fold more expensive. Trios will be analyzed within the same randomization arm (WGS or WES). This study is designed to quantify which acutely ill infants benefit from rapid genomic sequencing, by how much they benefit, how they benefit, which rapid genomic sequencing method is superior, and the cost effectiveness of such testing.

DETAILED DESCRIPTION:
Acutely ill infant inpatients who have an undiagnosed illness, and their families, will be eligible to participate in the study. The investigators will enroll up to 1,000 infants. Locally, the study population will be recruited from Rady Children's Hospital (RCH) inpatient population, primarily the neonatal intensive care unit (NICU), pediatric intensive care unit (PICU), and cardiovascular intensive care unit (CVICU), with a smaller population presenting to other hospital in-patient services. Recruitment will be targeted at the RCH main campus, but it may include referrals from satellite locations in the RCH network (particularly the RCH NICU network throughout San Diego County). All patients will continue to receive routine care as clinically indicated, including the state newborn screen and other genetic testing as determined by their treating providers. Half of the affected study participants will be randomized to receive rapid whole genome sequencing (WGS) and the other half will receive rapid whole exome sequencing (WES). Each arm will initially be analyzed using the patient's (proband's) sample only. If a proband-only analysis fails to yield a diagnosis, genomic data from the biological family members (typically parents), when available, will be used to supplement analysis (trio analysis). Occasionally, a second affected sibling may be available for family analysis. Not infrequently, the father is not available for study. Similarly, the investigators anticipate the need for targeted genetic analysis of biological parents, and possibly other family members, to confirm diagnostic results and/or provide additional information regarding inheritance.

The investigators anticipate that in rare cases a newborn may be so ill that the team lacks equipoise that the child can wait for the estimated ten day turnaround time of our send-out exome testing. In these rare cases, the PI, or his delegate, will decide if the child is not eligible for randomization. These children will remain in the research study throughout the entirety of the study, but will receive in-house ultra-rapid whole genome sequencing by the Rady Children's Institute for Genomic Medicine (RCIGM, also called RadyPGSMI) laboratory in lieu of either a rapid genome or rapid exome (both anticipated to be 10 day turn-arounds).

Enrollment will be sought within the first 96 hours following admission to RCH or an RCH network ICU or within 96 hours of meeting criteria for the study if the infant was not previously eligible. Patients and their family members who consent to participate will have their blood drawn and will be randomized to receive either rapid WGS or rapid WES. The initial symptom-driven analysis will be conducted on the patient's sample only (singleton analysis). If a diagnosis is not found promptly (within 24 hours) via a singleton analysis, the family (or any combination of parents and/or other family members) will be analyzed using the same technology that the patient was randomized to receive. Pathogenic and likely pathogenic variants (as determined by American College of Medical Genetics (ACMG) guidelines) that relate in part or in whole to the patient's current phenotype will be clinically confirmed and reported into the patients' medical record. Although the intention of the study is to return symptom-driven results to the medical record, the clinical report for confirmation of symptom-driven findings may include negative findings of testing. In the event that our analysis incidentally finds a pathogenic variant for which a treatment or intervention exists to improve morbidity and/or mortality, families may choose not to receive this additional information.

ELIGIBILITY:
Inclusion Criteria:

Individual in whom one of the following criteria is met:

1. Acutely ill inpatient of less than 4 months of age and within 96 hours of admission.
2. Acutely ill inpatient of less than 4 months of age and within 96 hours of development of an abnormal response to standard therapy for an underlying condition.
3. Acutely ill inpatient of less than 4 months of age and within 96 hours of development of clinical feature or laboratory test value suggestive of a genetic condition.
4. Biological relative of an infant enrolled in this study.

Exclusion Criteria:

Inpatients of greater than 4 months of age, or who do not meet any of the inclusion criteria, or with:

1. Neonatal infection or sepsis with normal response to therapy
2. Isolated prematurity
3. Isolated unconjugated hyperbilirubinemia
4. Hypoxic Ischemic Encephalopathy with clear precipitating event
5. Previously confirmed genetic diagnosis that explains their clinical condition (i.e. have a positive genetic test)
6. Isolated Transient Neonatal Tachypnea
7. Permission is unable to be obtained by a legal guardian or court-appointed representative within 96 hours of becoming eligible for enrollment.
8. Non-viable neonates - newborns less than 28 days of life with a modified code status (only full code patients may be enrolled).

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 213 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2024-07-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen F Kingsmore, MD, DSc, Principal Investigator — Rady Pediatric Genomics & Systems Medicine Institute
Locations (1):
- Rady Children's Institute for Genomic Medicine (RCIGM), San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Samples and data may be shared confidentially with collaborators, such as commercial laboratories or technology companies. All data and sample sharing will be strictly confidential. No identifying information will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication of results; Indefinitely
Access Criteria: Researchers must register at NBSTRN and request access to this dataset via the LPDR.
URL: https://nbstrn.org/

REFERENCES:
- [Background] Milko LV, Chen F, Chan K, Brower AM, Agrawal PB, Beggs AH, Berg JS, Brenner SE, Holm IA, Koenig BA, Parad RB, Powell CM, Kingsmore SF. FDA oversight of NSIGHT genomic research: the need for an integrated systems approach to regulation. NPJ Genom Med. 2019 Dec 10;4:32. doi: 10.1038/s41525-019-0105-8. eCollection 2019. PMID 31839987
- [Background] Kingsmore SF, Nofsinger R, Ellsworth K. Rapid genomic sequencing for genetic disease diagnosis and therapy in intensive care units: a review. NPJ Genom Med. 2024 Feb 27;9(1):17. doi: 10.1038/s41525-024-00404-0. PMID 38413639
- [Background] Chan K, Hu Z, Bush LW, Cope H, Holm IA, Kingsmore SF, Wilhelm K, Scharfe C, Brower A. NBSTRN Tools to Advance Newborn Screening Research and Support Newborn Screening Stakeholders. Int J Neonatal Screen. 2023 Oct 30;9(4):63. doi: 10.3390/ijns9040063. PMID 37987476
- [Background] Owen MJ, Lefebvre S, Hansen C, Kunard CM, Dimmock DP, Smith LD, Scharer G, Mardach R, Willis MJ, Feigenbaum A, Niemi AK, Ding Y, Van Der Kraan L, Ellsworth K, Guidugli L, Lajoie BR, McPhail TK, Mehtalia SS, Chau KK, Kwon YH, Zhu Z, Batalov S, Chowdhury S, Rego S, Perry J, Speziale M, Nespeca M, Wright MS, Reese MG, De La Vega FM, Azure J, Frise E, Rigby CS, White S, Hobbs CA, Gilmer S, Knight G, Oriol A, Lenberg J, Nahas SA, Perofsky K, Kim K, Carroll J, Coufal NG, Sanford E, Wigby K, Weir J, Thomson VS, Fraser L, Lazare SS, Shin YH, Grunenwald H, Lee R, Jones D, Tran D, Gross A, Daigle P, Case A, Lue M, Richardson JA, Reynders J, Defay T, Hall KP, Veeraraghavan N, Kingsmore SF. An automated 13.5 hour system for scalable diagnosis and acute management guidance for genetic diseases. Nat Commun. 2022 Jul 26;13(1):4057. doi: 10.1038/s41467-022-31446-6. PMID 35882841
- [Background] Kingsmore SF, Cole FS. The Role of Genome Sequencing in Neonatal Intensive Care Units. Annu Rev Genomics Hum Genet. 2022 Aug 31;23:427-448. doi: 10.1146/annurev-genom-120921-103442. Epub 2022 Jun 8. PMID 35676073
- [Result] Dimmock DP, Clark MM, Gaughran M, Cakici JA, Caylor SA, Clarke C, Feddock M, Chowdhury S, Salz L, Cheung C, Bird LM, Hobbs C, Wigby K, Farnaes L, Bloss CS, Kingsmore SF; RCIGM Investigators. An RCT of Rapid Genomic Sequencing among Seriously Ill Infants Results in High Clinical Utility, Changes in Management, and Low Perceived Harm. Am J Hum Genet. 2020 Nov 5;107(5):942-952. doi: 10.1016/j.ajhg.2020.10.003. PMID 33157007
- [Result] Cakici JA, Dimmock DP, Caylor SA, Gaughran M, Clarke C, Triplett C, Clark MM, Kingsmore SF, Bloss CS. A Prospective Study of Parental Perceptions of Rapid Whole-Genome and -Exome Sequencing among Seriously Ill Infants. Am J Hum Genet. 2020 Nov 5;107(5):953-962. doi: 10.1016/j.ajhg.2020.10.004. PMID 33157008
- [Result] Kingsmore SF, Cakici JA, Clark MM, Gaughran M, Feddock M, Batalov S, Bainbridge MN, Carroll J, Caylor SA, Clarke C, Ding Y, Ellsworth K, Farnaes L, Hildreth A, Hobbs C, James K, Kint CI, Lenberg J, Nahas S, Prince L, Reyes I, Salz L, Sanford E, Schols P, Sweeney N, Tokita M, Veeraraghavan N, Watkins K, Wigby K, Wong T, Chowdhury S, Wright MS, Dimmock D; RCIGM Investigators. A Randomized, Controlled Trial of the Analytic and Diagnostic Performance of Singleton and Trio, Rapid Genome and Exome Sequencing in Ill Infants. Am J Hum Genet. 2019 Oct 3;105(4):719-733. doi: 10.1016/j.ajhg.2019.08.009. Epub 2019 Sep 26. PMID 31564432
- [Result] Cakici JA, Dimmock D, Caylor S, Gaughran M, Clarke C, Triplett C, Clark MM, Kingsmore SF, Bloss CS. Assessing Diversity in Newborn Genomic Sequencing Research Recruitment: Race/Ethnicity and Primary Spoken Language Variation in Eligibility, Enrollment, and Reasons for Declining. Clin Ther. 2023 Aug;45(8):736-744. doi: 10.1016/j.clinthera.2023.06.014. Epub 2023 Jul 8. PMID 37429778
- [Result] Owen MJ, Batalov S, Ellsworth KA, Wright M, Breeding S, Hugh K, Kingsmore SF, Ding Y. Rapid Whole Genome Sequencing for Diagnosis of Single Locus Genetic Diseases in Critically Ill Children. Methods Mol Biol. 2023;2621:217-239. doi: 10.1007/978-1-0716-2950-5_12. PMID 37041447
- [Derived] Laurenzano SE, McFall C, Nguyen L, Savla D, Coufal NG, Wright MS, Tokita M, Dimmock D, Kingsmore SF, Newfield RS. Neonatal diabetes mellitus due to a novel variant in the INS gene. Cold Spring Harb Mol Case Stud. 2019 Aug 1;5(4):a004085. doi: 10.1101/mcs.a004085. Print 2019 Aug. PMID 31196892
- Available data/document: Individual Participant Data Set: 37114 — http://view.ncbi.nlm.nih.gov/dbgap-controlled
- Available data/document: Summary level phenotype data: 37114 — http://www.ncbi.nlm.nih.gov/projects/gap/cgi-bin/study.cgi?study_id=phs002094.v1.p1
- Available data/document: Subject Sample Telemetry Report (SSTR) for Subject and Sample IDs, consents, summary counts, processing status, and molecular and sequence sample uses: 37114 — http://www.ncbi.nlm.nih.gov/gap/sstr/report/phs002094.v1.p1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of acutely ill infants (age less than 1 year) during admission to the neonatal, pediatric or intensive care unit at Rady Children's Hospital, San Diego
Pre-assignment Details: Infants considered to be too severely ill at enrollment to be randomized to rapid diagnostic whole genome sequencing or rapid diagnostic whole exome sequencing were excluded from randomization and received ultra-rapid diagnostic whole genome sequencing with the fastest possible time to diagnosis.
Groups:
- Diagnostic Rapid Whole Genome Sequencing: Genetic test that looks at all coding and non-coding areas of the genome. Genomic sequencing and molecular diagnostic results.
- Diagnostic Rapid Whole Exome Sequencing: Genetic test that looks at all coding areas of the genome. Genomic sequencing and molecular diagnostic results.
- Ultra-rapid Diagnostic Whole Genome Sequencing: Infants considered to be too severely ill at enrollment to be randomized were excluded from randomization and received urWGS, with the fastest possible time to diagnosis.
Period: Overall Study
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing
Started | 94 | 95 | 24
Completed (Diagnostic report issued) | 94 | 95 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing | Total
Number analyzed (Participants) | 94 | 95 | 24 | 213
Age, Continuous [Median (Full Range); unit: Days] | 4 [1 to 105] | 5 [1 to 121] | 7.5 [2 to 67] | 5 [1 to 121]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 43 | 8 | 84
  Male | 61 | 52 | 16 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 42 | 10 | 88
  Not Hispanic or Latino | 57 | 52 | 14 | 123
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 6 | 2 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 2 | 5 | 0 | 7
  Black or African American | 3 | 2 | 1 | 6
  White | 58 | 55 | 17 | 130
  More than one race | 20 | 27 | 3 | 50
  Unknown or Not Reported | 5 | 4 | 2 | 11
Age at symptom onset [Median (Full Range); unit: Days] — Age in days. Participants are infants age less than 1 year who are admitted to a neonatal, pediatric, or cardiovascular intensive care unit for management of an acute illness. The age at symptom onset is the time between birth and onset of symptoms associated with the acute illness that led to their admission.
  Days | 0.4 [0 to 102] | 0.6 [0 to 120] | 3.1 [0 to 63] | 1 [0 to 120]

OUTCOME MEASURES:

1. Primary Outcome: Subject's Main Provider's Perceived Clinical Utility of Genomic Sequencing
Description: Perceived utility/benefit of sequencing based on "Clinician Assessment" questionnaire completed by patient's providers. Question: Was the test clinically useful? Response was measured on a 5-point Likert scale (very useful=5, useful=4, neutral=3, not very useful=2, not useful at all=1.
Time Frame: Within one week of the return of results
Population: Test perceived to be useful or very useful in "Clinician Assessment" questionnaire completed by patient's providers.
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing
Number analyzed (Participants) | 93 | 90 | 24
Participants | 66 | 66 | 24

2. Primary Outcome: Test Results Led to Change in Patient Management
Description: Test results led to Change in clinical management (select all that apply):
  * Surgical intervention added
  * Surgical intervention removed
  * Surgical intervention changed
  * Medication added
  * Medication removed
  * Medication changed
  * Diet changed
  * New specialty service sought
  * Prior specialty service no longer required
  * New imaging sought
  * Prior imaging cancelled
  * New test ordered
  * Prior testing cancelled
  * Screening for additional comorbidities added
  * Screening for additional comorbidities removed
  * Palliative care initiated
  * Palliative care withdrawn
  * Other: (text box for written description)
Time Frame: Within 1 week of return of results
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing
Number analyzed (Participants) | 93 | 90 | 24
Participants | 23 | 19 | 15

3. Primary Outcome: Test Led to Changes in Management That Altered Patient Outcome
Description: Primary physician perception of change in outcome
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing
Number analyzed (Participants) | 93 | 90 | 24
Participants | 9 | 17 | 6

4. Secondary Outcome: Diagnostic Proportion for Whole Genome Sequencing (WGS) and Whole Exome Sequencing (WES)
Description: WGS and WES are two clinical diagnostic test modalities. Results of testing were placed in the electronic medical record. Results either provided a molecular diagnosis that explained the patient's condition or did not. The diagnostic proportion is the number of patients who received a molecular diagnosis by the test modality divided by the total number of patients who were tested by that modality.
Time Frame: Within approximately 30 days of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing
Number analyzed (Participants) | 94 | 95 | 24
Participants | 18 | 19 | 11

5. Secondary Outcome: Result Within 7 Days of Sample Receipt
Description: Time to result.
Time Frame: Within 7 days of sample receipt
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing
Number analyzed (Participants) | 94 | 95 | 24
Participants | 10 | 4 | 17

6. Secondary Outcome: Parental Perceived Usefulness of Test
Description: Parental perception that test was useful
Time Frame: Within one week of the return of results and approximately one year after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing
Number analyzed (Participants) | 70 | 71 | 20
Participants | 54 | 55 | 15

7. Secondary Outcome: Parental Perception of Test Benefit for Their Infant
Description: Parental perception that the test benefitted their infant
Time Frame: Within one week of the return of results and approximately one year after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing
Number analyzed (Participants) | 70 | 71 | 20
Participants | 58 | 50 | 13

8. Secondary Outcome: Parental Decisional Regret With Sequencing
Description: Markers of harm in genetic diagnosis as evidenced by Brehaut's Decisional Regret scale. Scale 0-100. Higher scores indicate higher regret.
Time Frame: Within one week of the return of results and approximately one year after enrollment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing
Number analyzed (Participants) | 70 | 71 | 20
score on a scale | 5 [0 to 60] | 0 [0 to 100] | 15 [0 to 30]

ADVERSE EVENTS:
Time Frame: 1 year for parental perception of harm; 28 days for mortality
Description: Adverse event measured was parental perception that test was harmful to infant. 28-day mortality was a demographic measure of the severity of illness of patients. 28-day mortality not due to testing but rather to underlying disease.
Arm/Group | Diagnostic Rapid Whole Genome Sequencing | Diagnostic Rapid Whole Exome Sequencing | Ultra-rapid Diagnostic Whole Genome Sequencing
All-Cause Mortality (participants affected / at risk) | 0/94 | 3/95 | 5/24
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/95 | 0/24
Other Adverse Events (participants affected / at risk) | 0/94 | 3/95 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diagnostic Rapid Whole Genome Sequencing (N=94) | Diagnostic Rapid Whole Exome Sequencing (N=95) | Ultra-rapid Diagnostic Whole Genome Sequencing (N=24)
Parental perception that test was harmful to infant (Social circumstances) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT03211039/Prot_SAP_000.pdf